CLINICAL TRIAL: NCT01380821
Title: DNA Double-strand Breaks Following Myocardial Scintigraphy
Brief Title: DNA Double-strand Breaks After SPECT
Acronym: DSB-SPECT
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Marc Dewey, Charité
Other Study IDs: EA4/004/11
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
Keywords: clinical indication for myocardial SPECT; suspected or known coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPECT: Patients clinically indicated to undergo myocardial SPECT in our institution.
  Interventions: Radiation: Myocardial SPECT

INTERVENTIONS:
Radiation: Myocardial SPECT — Myocardial SPECT according to clinical standards for patients with a clinical indication to undergo this imaging test.

SUMMARY:
Ionizing radiation has a number of harmful effects in humans. The most important among these is the induction of cancer. It is assumed that damage to DNA in the nucleus of a single cell can induce cancer. Among the different types of lesions inducted, DNA double-strand breaks (DSBs) are considered to be the most relevant effects that can initiate carcinogenesis.

The investigators are already conducting several other studies to prospectively compare the inducted DSBs by coronary CT-angiography and conventional coronary angiography. Extending these examinations to investigate the induced DSBs by myocardial scintigraphy allows a comparison of all three relevant imaging methods of the heart that incorporate ionizing radiation.

To evaluate this, the investigators are planning to examine patients who are scheduled for a clinically indicated myocardial scintigraphy. These examinations are routinely done by the Department of Nuclear Medicine in either a 1-day or a 2-day protocol according to the diagnostic reference values of the Federal Department for Radiological Protection. Blood samples will be taken from these patients at predefined time steps before and after the examination and DNA double-strand breaks will be determined from these blood samples specifically considering the applied activity of the tracer and the exposition kinetics.

ELIGIBILITY:
Inclusion Criteria:

* myocardial SPECT clinically indicated

Exclusion Criteria:

* acute leukaemia or lymphoma
* radiation or chemotherapy in the last 6 months
* x-ray or scintigraphy within the last 3 days
* age below 18 years
* eGFR of below 60 ml/min

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients clinically indicated to undergo myocardial SPECT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Radiation-induced DNA double-strand breaks after myocardial scintigraphy. | 48 hours
  DNA double-strand breaks will be measured before and up to 48 hours after radiation.

SECONDARY OUTCOMES:
Comparison of radiation-induced DSBs with activity used for myocardial scintigraphy. | Activity will be measured 5 min and 1h after injection of the technetium tracer for SPECT.
  DNA double-strand breaks will be compared with injected activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Geisel D, Heverhagen JT, Kalinowski M, Wagner HJ. DNA double-strand breaks after percutaneous transluminal angioplasty. Radiology. 2008 Sep;248(3):852-9. doi: 10.1148/radiol.2483071686. PMID 18710979